CLINICAL TRIAL: NCT03910556
Title: Predictive Factors of Re-craniotomy and Major Non-neurological Complications in Elective Neurosurgery: A Prospective Cohort Study
Brief Title: Re-craniotomy and Complications After Elective Neurosurgery
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Collaborators: Yodying Punjasawadwong (Unknown); Prangmalee Leucharussamee (Unknown); Ananchanok Saringkarinkul (Unknown); Patipan Krungsri (Unknown)
Responsible Party: Principal Investigator, Pathomporn Pin on, M.D., Assistant Professor, Chiang Mai University
Other Study IDs: ANE-2561-05961
Record Dates: First submitted 2019-04-06; First posted 2019-04-10 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Brain Tumor; Brain Metastases; Brain Cancer; Brain Neoplasms
Keywords: re-craniotomy; major non-neurological complications; neurosurgery; brain tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Propofol; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no complication: the patients who did not develop any kind of complication and no re-craniotomy
  Interventions: Drug: Propofol
- with complication (s): the patients who developed at least one of non-neurological complication or required re-craniotomy
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — intraoperative factors
  Other Names: surgical duration; operation; blood loss; blood used; fluid volume administration

SUMMARY:
This study is a prospective cohort study to find the incidence of re-craniotomy and predictive factors. The secondary outcomes are to find the incidence of major non-neurological complications and predictive factors.

DETAILED DESCRIPTION:
Demographic data include age, gender, preoperative neurological assessment, diagnosis, operation, surgical position, ASA physical status, dexamethasone requirement, anticonvulsant therapy, airway assessment, and blood component reservation.

Intraoperative information contain anesthetic technique, total dosage of propofol, fentanyl, and other anesthetic agents, total blood loss, types and amount of fluid replacement, volume of blood transfusion, latest body temperature, and the ability of safe extubation.

Postoperative complications will be categorized in to general conditions, neurological complications, and systemic problems. General conditions such as on endotracheal tube overnight and postoperative blood transfusion. Neurological complications include worsen increased ICP, intracranial hematoma, seizures, newly-developed motor deficit, cranial nerve palsy, CSF rhinorrhea, and emergency re-craniotomy. Systemic problems are hypothermia, electrolyte imbalance, anemia, hypertension, and hyperglycemia. Postoperative nausea and vomiting and the rescued anti-emetic drugs will be recorded. Postoperative anti-epileptic drug (AED) and pain medication will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for elective craniotomy during 2017-2019
* Patients who are planned for general anesthesia
* Patients have read the study information and signed in the consent form

Exclusion Criteria:

* Patients who are unable to understand and sign in the consent form
* Patients who are scheduled for minor surgical procedures such as ventriculostomy and VP-shunt

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The adult patients who were scheduled for craniotomy to remove tumor
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
re-craniotomy | the first 24 hours
  number of participants who required re-craniotomy assessed by the neurosurgeon
predictive factors of re-craniotomy | the first 24 hours
  types of perioperative factors to predict the occurrence of re-craniotomy

SECONDARY OUTCOMES:
incidence of major non-neurological complications | the first 24 hours
  number of participants who develop any major systemic complications
predictive factors of major non-neurological complications | the first 24 hours
  types of predictive factors to predict the occurrence of major non-neurological complications

CONTACTS AND LOCATIONS:
Overall Officials: Pathomporn Pin-on, MD, Principal Investigator — Chiang Mai University

IPD SHARING:
Plan to Share IPD: No